CLINICAL TRIAL: NCT00633191
Title: Post Marketing Study of Anti-pseudomonas IgY in Prevention of Recurrence of Pseudomonas Aeruginosa Infections Infections in Cystic Fibrosis (CF) Patients
Brief Title: Anti-pseudomonas IgY to Prevent Infections in Cystic Fibrosis
Acronym: PseudIgY
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Immunsystem AB (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pseud-IgY-1
Record Dates: First submitted 2008-03-04; First posted 2008-03-11 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Cystic Fibrosis; Infection; Pseudomonas Aeruginosa
Keywords: Cystic fibrosis; Prevention; Infection; Pseudomonas aeruginosa; Gargle
MeSH Terms: conditions — Cystic Fibrosis; Infections; Pseudomonas Infections | interventions — Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Anti-pseudomonas IgY gargle (Experimental): Intervention: Gargles with anti-pseudomonas IgY every night
  Interventions: Drug: Anti-pseudomonas IgY gargle

INTERVENTIONS:
Drug: Anti-pseudomonas IgY gargle — Gargle (solution), > 5FKU, every night after toothbrushing, life-long
  Other Names: oral immunotherapy; Yolk antiboidies

SUMMARY:
Hypothesis: Daily gargling with specific avian antibodies against Pseudomonas aeruginosa will prevent infections with this bacteria in patients with Cystic fibrosis (CF).

DETAILED DESCRIPTION:
"Anti-pseudomonas IgY" is prepared from eggs of hens that have been vaccinated with Pseudomonas aeruginosa. The hens farm is under veterinary control according to Swedish rules. The drug is prepared with a water dilution method according to GMP standards (approved by Swedish MPA). Patients with CF who are intermittently but not chronically infected with P. aeruginosa get a short course of antibiotics to eradicate the bacteria. Thereafter they start to gargle with a solution of "anti-pseudomonas IgY" every night to prevent a new infection. Preliminary results have shown that it takes a significantly longer time to get a new infection and that the patients get fewer infections than control patients. In addition, results tentatively indicate that: patients have not got any new opportunistic bacteria or fungi (B. Cepacia, S. Maltophilia, A. Xylosoxidans, atypical Mycobacteria, Aspergillus Fumigatus); that use of antibiotics is greatly diminished; that the lung functions and nutritional conditions are maintained.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of cystic fibrosis
* Colonized with Pseudomonas aeruginosa
* informed consent

Exclusion Criteria:

* Egg allergy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2003-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Sputum culture positive for Pseudomonas aeruginosa | Prospective

SECONDARY OUTCOMES:
Pulmonary function | Prospective

CONTACTS AND LOCATIONS:
Overall Officials: Annika Hollsing, MD, PhD, Principal Investigator — Uppsala Children´s University Hospital
Locations (1):
- Cystic fibrosis centre,Children´s University Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carlander D, Kollberg H, Larsson A. Retention of specific yolk IgY in the human oral cavity. BioDrugs. 2002;16(6):433-7. doi: 10.2165/00063030-200216060-00004. PMID 12463766
- [Background] Kollberg H, Carlander D, Olesen H, Wejaker PE, Johannesson M, Larsson A. Oral administration of specific yolk antibodies (IgY) may prevent Pseudomonas aeruginosa infections in patients with cystic fibrosis: a phase I feasibility study. Pediatr Pulmonol. 2003 Jun;35(6):433-40. doi: 10.1002/ppul.10290. PMID 12746939
- [Background] Nilsson E, Kollberg H, Johannesson M, Wejaker PE, Carlander D, Larsson A. More than 10 years' continuous oral treatment with specific immunoglobulin Y for the prevention of Pseudomonas aeruginosa infections: a case report. J Med Food. 2007 Jun;10(2):375-8. doi: 10.1089/jmf.2006.214. PMID 17651078
- [Background] Nilsson E, Larsson A, Olesen HV, Wejaker PE, Kollberg H. Good effect of IgY against Pseudomonas aeruginosa infections in cystic fibrosis patients. Pediatr Pulmonol. 2008 Sep;43(9):892-9. doi: 10.1002/ppul.20875. PMID 18680179
- [Background] Nilsson E, Amini A, Wretlind B, Larsson A. Pseudomonas aeruginosa infections are prevented in cystic fibrosis patients by avian antibodies binding Pseudomonas aeruginosa flagellin. J Chromatogr B Analyt Technol Biomed Life Sci. 2007 Sep 1;856(1-2):75-80. doi: 10.1016/j.jchromb.2007.05.029. Epub 2007 Jun 2. PMID 17581799
- [Background] Nilsson E, Hanrieder J, Bergquist J, Larsson A. Proteomic characterization of IgY preparations purified with a water dilution method. J Agric Food Chem. 2008 Dec 24;56(24):11638-42. doi: 10.1021/jf802626t. PMID 19053374
- [Background] Nilsson E, Stalberg J, Larsson A. IgY stability in eggs stored at room temperature or at +4 degrees C. Br Poult Sci. 2012;53(1):42-6. doi: 10.1080/00071668.2011.646951. PMID 22404803
- [Derived] Hurley MN, Smith S, Forrester DL, Smyth AR. Antibiotic adjuvant therapy for pulmonary infection in cystic fibrosis. Cochrane Database Syst Rev. 2020 Jul 16;7(7):CD008037. doi: 10.1002/14651858.CD008037.pub4. PMID 32671834